CLINICAL TRIAL: NCT06339086
Title: A Multicenter, Randomized, Open-label and Parallel-controlled Phase III Study to Compare the Efficacy and Safety of Semaglutide Injection With Ozempic® in the Treatment of Type 2 Diabetes Subjects With Poor Glycemic Control on Metformin
Brief Title: Efficacy and Safety of Semaglutide Injection in Subjects With Type 2 Diabetes
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chengdu Brilliant Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BPR-201-I-III-01
Record Dates: First submitted 2024-03-18; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide; Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Semaglutide Injection (Experimental): Semaglutide 0.25mg、0.5mg、1.0mg
  Metformin ≥ 1500mg/day (or maximum tolerated dose ≥ 1000mg/day) and ≤2000mg/day
  Interventions: Drug: Semaglutide Injection; Drug: Metformin
- Ozempic® (Active Comparator): Ozempic® 0.25mg、0.5mg、1.0mg
  Metformin ≥ 1500mg/day (or maximum tolerated dose ≥ 1000mg/day) and ≤2000mg/day.
  Interventions: Drug: Semaglutide Injection(Ozempic®); Drug: Metformin

INTERVENTIONS:
Drug: Semaglutide Injection — The subject will receive either a dose of semaglutide subcutaneously once weekly. The initial dose of semaglutide is 0.25mg per week and will be increased to 0.5mg after 4 weeks. After 4 weeks of 0.5mg administration, the dose will be increased to 1mg and continued at a stable does of 1mg for 24 weeks.
  Treatment duration 32 weeks.
  Arms: Semaglutide Injection
Drug: Semaglutide Injection(Ozempic®) — The subject will receive either a dose of Ozempic® subcutaneously once weekly. The initial dose of semaglutide is 0.25mg per week and will be increased to 0.5mg after 4 weeks. After 4 weeks of 0.5mg administration, the dose will be increased to 1mg and continued at a stable does of 1mg for 24 weeks.
  Treatment duration 32 weeks.
  Other Names: Ozempic®
  Arms: Ozempic®
Drug: Metformin — Metformin ≥ 1500mg/day (or maximum tolerated dose ≥ 1000mg/day) and ≤2000mg/day.
  Treatment duration 32 weeks.
  Other Names: Glucophage®

SUMMARY:
The goal of this clinical trial is to evaluate the similarities in efficacy and safety of semaglutide injection and Ozempic® in patients with type 2 diabetes who have poor glycemic control after metformin treatment.

Participants will receive either a dose of semaglutide or Ozempic® once weekly (subcutaneous injection) as add-on to metformin for 32 weeks.

Researchers will compare the outcomes of semaglutide and Ozempic® group to see if the efficacy, safety, pharmacokinetics, and immunogenicity of them are similar.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in this study, be able to communicate well with the investigator, understand and voluntarily complete the research process in accordance with this protocol, and sign the Informed Consent Form (ICF).
2. Male or female, aged ≥18 and ≤75 years old at the time of signing the ICF.
3. Diagnosis of type 2 diabetes for at least 6 months (WHO, 1999) at screening.
4. Use a stable dose of metformin for at least 60 days before screening (stable dose of metformin: ≥1500 mg/day or maximum tolerated dose ≥1000 mg/day).
5. Glycosylated Hemoglobin(HbA1c) >7.0% and <11.0% at screening (local lab).
6. BMI ≥18.5 and ≤35 kg/m2 at screening.

Exclusion Criteria:

1. Laboratory tests meeting any of the following criteria at screening:

   1. Calcitonin ≥50ng/L (pg/mL);
   2. Blood amylase ≥3×ULN (upper limit of normal value);
   3. Blood lipase ≥3×ULN;
   4. Triglycerides ≥5.7mmol/L (500mg/dL);
   5. Alanine aminotransferase ≥3×ULN;
   6. Aspartate aminotransferase ≥3×ULN;
   7. Total bilirubin ≥2×ULN;
   8. Estimated glomerular filtration rate (eGFR) <60ml/min/1.73m2 (eGFR=175×Scr-1.234 (mg/dl)×age-0.179 (female×0.79), Scr unit conversion: 1mg/dl = 88.4μmol/L).
2. Positive HIV antibodies at screening.
3. Patients who have received other anti-diabetic drugs other than metformin within 60 days before screening. Such drugs include, but are not limited to, alpha-glycosidase inhibitors (such as acarbose), thiazolidinediones, glucagon-like peptide-1(GLP-1) analogs, dipeptidyl peptidase 4 (DPP-4) inhibitors, except short-term treatment with insulin (cumulative insulin treatment is allowed for ≤7 days within 60 days before screening).
4. Patients who have used GLP-1 receptor agonists within 3 months before screening, or have stopped using GLP-1 receptor agonists due to poor safety or efficacy.
5. Patients who have used weight loss drugs or have a weight change of more than 5% within 3 months before screening.
6. Continuous or cumulative use of systemic glucocorticoids for more than 7 days within 3 months before screening (systemic glucocorticoids: intravenous, oral or intra-articular glucocorticoid treatment).
7. Plan to receive glucocorticoids, immunosuppressants, or other drugs (except topical medications and inhaled preparations) that are assessed as unsuitable during the trial by the investigator.
8. Those who have participated in other clinical trials and received experimental drugs or placebo intervention within 3 months before screening (except those who only signed the ICF and did not receive any drug or placebo).
9. Those who are known to be allergic to the investigational drug or its excipients, or have a history of allergy to GLP-1 drugs, or are in an allergic state at the time of screening, or are unfit for the study due to allergy risks, per investigator's judgment.
10. Diagnosis of type 1 diabetes, diabetes caused by pancreatogenic injury or other special types of diabetes.
11. Have a history of acute diabetic complications (diabetic ketoacidosis, lactic acidosis or hyperosmolar hyperglycemic state) within 6 months before screening.
12. Recurrent (≥3 times) severe hypoglycemia or asymptomatic hypoglycemia events within 6 months before screening.
13. Patients who have hemoglobinopathies or hemolytic anemia, have received blood or plasma products within 3 months before screening, or have donated blood or lost more than 400 mL of blood within 3 months before screening.
14. History of congestive heart failure: New York Heart Association (NYHA) Class IV.
15. Patients who have acute coronary syndrome or cerebrovascular event (except old lacunar infarction) within 3 months before screening, including but not limited to acute myocardial infarction, unstable angina, stroke/transient cerebral ischemia attack, or have undergone heart-related surgery (including coronary artery bypass grafting, percutaneous coronary intervention) within 3 months before screening, or have poor blood pressure control at the time of screening (defined as systolic blood pressure ≥160 millimeter of mercury(mmHg) and /or diastolic blood pressure ≥100 mmHg with antihypertensive drugs) or any other cardiovascular/cerebrovascular diseases that are not suitable for participating in this trial.
16. History of proliferative retinopathy or diabetic macular edema, or any other unstable retinopathy (rapidly progressive) recorded in medical history and may require treatment during the study.
17. Patients with a history of acute/chronic pancreatitis, symptomatic gallbladder (such as multiple gallbladder stones, excluding cholecystectomy), pancreatic injury, or other conditions that may lead to high risk for pancreatitis.
18. Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN2).
19. Diagnosis of malignant tumors within 5 years before screening (except for adequately treated cervical carcinoma in situ, basal cell or squamous cell skin cancer).
20. Patients who have clinically significant gastric emptying abnormalities (such as severe diabetic gastroparesis, gastric outlet obstruction, etc.), have undergone or plan to undergo surgery that affects gastric emptying during the study period, or have long-term use of drugs that affect gastrointestinal motility.
21. Patients with history of alcohol abuse or drug addiction within 6 months before screening; or who have a mental illness (such as depression, etc.) that the may affect participation in the study, in the judgment of the Investigator.
22. Uncured active or recurrent bacterial, fungal or viral infection before randomization.
23. Females who are pregnant or lactating, or have a positive pregnancy test (woman of childbearing potential).
24. During the trial, men and women who have plans to have children or are of childbearing potential but not willing to use effective contraceptive methods.
25. In the judgment of the investigator, the patient suffers from diseases that may endanger his or her safety or compliance with the protocol, or other conditions that are not suitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | Week 32
  Change from baseline to week 32 in Glycosylated Hemoglobin(HbA1c).

SECONDARY OUTCOMES:
Change in HbA1c | Week 20
  Change from baseline to week 20 in HbA1c.
Change in FPG | Week 20，32
  Change from baseline to week 20, 32 in Fasting Plasma Glucose(FPG).
Proportion of participants who achieved HbA1c<7.0%，HbA1c≤6.5% | Week 20，32
  Proportion of participants who achieved HbA1c<7.0%，HbA1c≤6.5% at week 20, 32.
Proportion of participants who achieved HbA1c<7.0%，HbA1c≤6.5% with no hypoglycemic event | Week 20，32
  Proportion of participants who achieved HbA1c<7.0%，HbA1c≤6.5% with no confirmed symptomatic hypoglycemic event reported after treatment.
Change in Body Weight | Week 20，32
  Change from baseline to week 20, 32 in Body Weight.
Proportion of participants with Weight Loss≥5%, ≥10% and ≥15% | Week 20，32
  Proportion of participants with Weight Loss≥5%, ≥10% and ≥15% at week 20, 32.
Change in Diastolic and Systolic Blood Pressure | Week 32
  Change from baseline to week 32 in Diastolic and Systolic Blood Pressure.
Changes in Blood Lipids | Week 32
  Changes baseline to week 32 in Blood Lipids: Total Cholesterol, Low-density Lipoprotein Cholesterol, High-Density Lipoprotein Cholesterol, and Triglycerides.
Incidence and severity of Adverse Events | Week 32
  Incidence and severity of Adverse Events during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Dalong Zhu, PhD, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School

IPD SHARING:
Plan to Share IPD: No